CLINICAL TRIAL: NCT05863858
Title: High Eradication Rate of Helicobacter Pylori Infection With Moxifloxacin-Based Triple Therapy in Comparison With Levofloxacin-Based Sequential Therapy: Randomized Controlled Trials
Brief Title: Eradication of H. Pylori Infection With Moxifloxacin
Acronym: RCT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Iyad Naeem Muhammad, PhD (Other)
Responsible Party: Sponsor-Investigator, Iyad Naeem Muhammad, PhD, Associate Professor, University of Karachi
Organization: University of Karachi (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RCT-HP-01
Record Dates: First submitted 2023-03-25; First posted 2023-05-18 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Helicobacter Pylori Infection; Helicobacter Pylori Infection, Susceptibility to
Keywords: Triple therapy with moxifloxacin; Helicobacter pylori; Levofloxacin sequential therapy; Stool Antigen test
MeSH Terms: interventions — BID protein, human; Omeprazole; Tinidazole; Levofloxacin; Amoxicillin; Moxifloxacin

STUDY DESIGN:
Intervention Model Description: Patients were randomized into two regimens:
  1. Levofloxacin 500mg BID, Amoxicillin 1 gm BID, Omeprazole 20 mg BID for first five days followed by Levofloxacin 500 mg BID, Tinidazole 500mg BID, Omeprazole 20 mg BID, or
  2. Moxifloxacin 400 mg OD, Amoxicillin 1 gm BID, Omeprazole 20 mg BID.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Levofloxacin-based sequential Therapy (Active Comparator): 1. Tablets Levofloxacin 500mg BID for the first five days
  2. Tablet Amoxicillin 1 gm BID for first five days
  3. Capsules Omeprazole 20 mg BID for first five days followed by
  1. Tablet Levofloxacin 500 mg BID for five days 2. Tablet Tinidazole 500mg BID for five days 3. Capsule Omeprazole 20 mg BID for five days
  Infection eradication will be observed and confirmed by stool antigen test correlated with the signs and symptoms
  Interventions: Drug: Sequential Regimen: Levofloxacin 500 mg BID, Amoxicillin 1 gm BID, omeprazole 20 mg BID for first five days followed by Levofloxacin 500 mgBID, Tinidazole 500 mg BID, Omeprazole 20 mg BID
- Moxifloxacin-based Triple Therapy (Active Comparator): 1. Tablet Moxifloxacin 400 mg OD for ten days
  2. Tablet Amoxicillin 1 gm BID for ten days
  3. Capsule Omeprazole 20 mg BID for ten days
  Infection eradication will be observed and confirmed with a stool antigen test along with patient compliance and tolerability observance.
  Interventions: Drug: Triple Regimen: Moxifloxacin 400mg OD, Amoxicillin 1 gm BID, Omeprazole 20mgBID

INTERVENTIONS:
Drug: Sequential Regimen: Levofloxacin 500 mg BID, Amoxicillin 1 gm BID, omeprazole 20 mg BID for first five days followed by Levofloxacin 500 mgBID, Tinidazole 500 mg BID, Omeprazole 20 mg BID — The eradication rate of H. Pylori with levofloxacin-based sequential therapy
  Other Names: Levofloxacin; Amoxicillin; Omeprazole; Tinidazole
  Arms: Levofloxacin-based sequential Therapy
Drug: Triple Regimen: Moxifloxacin 400mg OD, Amoxicillin 1 gm BID, Omeprazole 20mgBID — The eradication rate of H. Pylori with moxifloxacin-based triple therapy
  Other Names: Moxifloxacin; Amoxicillin; Omeprazole
  Arms: Moxifloxacin-based Triple Therapy

SUMMARY:
The main objective of the study is to compare the effectiveness of moxifloxacin triple therapy with levofloxacin-based sequential therapy in terms of eradication rate, safety, and patient compliance.

DETAILED DESCRIPTION:
Patients who were confirmed to be positive for Helicobacter Pylori infection were randomly assigned to the eradication treatments. At four weeks after completion of eradication therapy, H. pylori tests were performed with a Stool antigen test.

ELIGIBILITY:
Inclusion Criteria:

1. Successful isolation of H. pylori from the patient, and
2. patients of at least 18 years of age.

Exclusion Criteria:

1. age under 18 years
2. presence of clinically signiﬁcant associated conditions (insulin-dependent diabetes mellitus, gastrointestinal bleeding, neoplastic diseases, coagulation disorders, and neurologic, metabolic, hematological or endocrine hepatic, cardiorespiratory, or renal diseases),
3. previous gastric surgery,
4. allergy to any of the drugs used in the study, and (5) pregnancy or breastfeeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-06-08 (Actual)

PRIMARY OUTCOMES:
Helicobacter pylori status one month after treatment. | One month after finishing with therapy.
  Helicobacter pylori status (positive or negative), will be measured by stool test, one month after finishing with therapy.

SECONDARY OUTCOMES:
Compliance of patients in both therapy groups in treatment of Helicobacter pylori infection. | One month after finishing with therapy.
  Compliance will be measured by counting pills that were taken during therapy. More than or equal 80 % of taken pills will be consider as good compliance
Adverse effects of therapy in both groups in treatment of Helicobacter pylori infection. | One month after finishing with therapy.
  Patients will be asked to report any adverse effect that occurred during treatment. They will be divided into groups according to the degree of limiting daily activities: no adverse effects; mild (no limit of activities); moderate (partially limited activities); severe (completely limited activities).

CONTACTS AND LOCATIONS:
Overall Officials: Iyad N Muhammad, Ph.D., Principal Investigator — Faculty of Pharmacy and Pharmaceutical Sciences, University of Karachi
Locations (1):
- Jamal Noor Hospital, Karachi, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared and made available for other researchers after due coding. The data will be summarized and tabulated in the thesis and article manuscripts. The IPD would include the basic information and demographic data, the treatment protocols, informed consent, and the outcome measures data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: The data will be shared and made permanently available on the formats mentioned above by January 2024.
Access Criteria: The data will be shared by the researches in RCT, working on H. pylori therapy or diagnosis. Communication would be electronically made through emails.

REFERENCES:
- [Background] Rakici H, Ayaz T, Akdogan RA, Bedir R. Comparison of levofloxacin- and moxifloxacin-based triple therapies with standard treatment in eradication of Helicobacter pylori as first-line therapy. Digestion. 2014;90(4):261-4. doi: 10.1159/000369788. Epub 2014 Dec 24. PMID 25547786
- [Background] Mori H, Suzuki H. Update on quinolone-containing rescue therapies for Helicobacter pylori infection. World J Gastroenterol. 2020 Apr 21;26(15):1733-1744. doi: 10.3748/wjg.v26.i15.1733. PMID 32351290
- [Background] Hsu PI, Tsay FW, Kao JY, Peng NJ, Chen YH, Tang SY, Kuo CH, Kao SS, Wang HM, Wu IT, Shie CB, Chuah SK, Wu DC; Taiwan Acid-related Disease, Microbiota (TARD-M) Consortium. Tetracycline-levofloxacin versus amoxicillin-levofloxacin quadruple therapies in the second-line treatment of Helicobacter pylori infection. Helicobacter. 2021 Oct;26(5):e12840. doi: 10.1111/hel.12840. Epub 2021 Aug 12. PMID 34390083
- [Background] Hwang JJ, Lee DH, Yoon H, Shin CM, Park YS, Kim N. Efficacy of moxifloxacin-based sequential and hybrid therapy for first-line Helicobacter pylori eradication. World J Gastroenterol. 2015 Sep 21;21(35):10234-41. doi: 10.3748/wjg.v21.i35.10234. PMID 26401089